CLINICAL TRIAL: NCT03822052
Title: A Randomized Controlled Trial Comparing D5LR to LR for Induction of Labor and Time to Delivery in Multiparous and Primiparous Patient's With Favorable and Unfavorable Bishop's Scores
Brief Title: The Use of D5LR Versus LR for Induction of Labor and Time to Delivery in Multiparous and Primiparous Patient's With Favorable and Unfavorable Bishop's Scores
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascension Health (Industry)
Responsible Party: Principal Investigator, Katelyn Hartung, DO, Postgraduate Year 3, Ascension Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ME 19 004
Record Dates: First submitted 2019-01-18; First posted 2019-01-30 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Induction of Labor Affected Fetus / Newborn
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Primiparous Patient, Unfavorable Bishop Score (Active Comparator): Patient to receive D5LR or LR at 125 cc/hr
  Interventions: Other: Lactated ringers; Other: 5% dextrose lactated ringers
- Primiparous Patient, Favorable Bishop Score (Active Comparator): Patient to receive D5LR or LR at 125 cc/hr
  Interventions: Other: Lactated ringers; Other: 5% dextrose lactated ringers
- Multiparous patient, Unfavorable Bishop Score (Active Comparator): Patient to receive D5LR or LR at 125 cc/hr
  Interventions: Other: Lactated ringers; Other: 5% dextrose lactated ringers
- Multiparous patient, Favorable Bishop Score (Active Comparator): Patient to receive D5LR or LR at 125 cc/hr
  Interventions: Other: Lactated ringers; Other: 5% dextrose lactated ringers

INTERVENTIONS:
Other: Lactated ringers — IV fluid
Other: 5% dextrose lactated ringers — IV fluid

SUMMARY:
Currently, the optimum IV fluid for induction of labor is unknown. The goal of this study is to determine the optimum fluid for induction of labor, D5LR versus LR. The investigators hypothesize that patients assigned to the D5LR group will have a shorter induction of labor when compared to patient's in the LR group.

DETAILED DESCRIPTION:
Induction of labor is increasingly common in the United States, as the overall rate has increased from 9.5% in 1990 to 22.1% in 2006 with the goal to stimulate contractions prior to the onset of spontaneous labor. Cesarean delivery rates are also at an all-time high in the U.S., with more than 32% of patients being delivered by Cesarean in 2009. One of the most common indications for Cesarean section is a prolonged labor course. Patient's with a prolonged labor course are also at risk for infections, including chorioamnionitis and endometritis, as well as an increased risk of postpartum hemorrhage. There is a lack of information on ways to help shorten labor to potentially minimize these risks.

The uterus is comprised of skeletal muscle, and labor has been likened to prolonged rigorous exercise. While oral hydration has been endorsed by ACOG for low-risk women in spontaneous labor, solid foods should be avoided. In turn, women with a prolonged induction or labor may benefit from glucose supplementation via IV fluids.

The DEXTRONS study, J. Pare et al., looked at supplementation of D5LR versus normal saline in nulliparous patients who presented for a favorable induction of labor. This study showed a significant reduction in active labor time in the D5LR group versus the normal saline group.

Currently, at Genesys Regional Medical Center, lactated ringers is the preferred IV fluid for patients presenting for induction of labor. This study will randomly assign patients to D5LR versus lactated ringers and examine the length of time from induction to delivery to determine if glucose supplementation has an effect on reducing length of induction in both nulliparous and multiparous patients for either a favorable induction of labor or an induction for post-dates. Secondary outcomes will include Apgar scores, need for special care nursery/NICU admissions, and mode of delivery. The study will begin in January 2019 and continue through July 2019. Patients who presented to labor and delivery and consent to be included in the study will be randomized to each group.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women, age 18 - 45, that were admitted for induction of labor without any co-morbid conditions and their respective newborns with
* Induction of labor
* Singleton pregnancies
* Vertex presentation
* Pregnancies at 39 0/7 weeks gestation - 41 6/7 weeks gestation
* All races/ethnicities

Exclusion Criteria:

* Multifetal gestations
* Noncephalic presentation
* Preexisting medical conditions:
* Maternal cardiac disease
* Lung diseases
* Chronic hypertension
* Pregestational or gestational diabetes
* gHTN or Pre-Eclampsia
* medical indication for induction of labor (olighydramnios, IUGR)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Time of induction | 492 min +/- 35 min
  Time from start of labor induction to delivery of infant

SECONDARY OUTCOMES:
Time of Active Labor | 4 hours +/- 3 hours
  time from 6 cm dilation until delivery of infant
Apgar Scores | 492 min +/- 35 min
  validated measure of infant health
Mode of Delivery | 492 min +/- 35 min
  Cesarean section vs SVD vs OVD
Neonatal ICU admissions | 24 hours after delivery
  ICU or special care nursery admissions
Need for respiratory support | 24 hours after delivery
  Neonatal need for respiratory support
Transfer to tertiary care center | 24 hours after delivery
  neonatal need for transfer to higher level NICU

CONTACTS AND LOCATIONS:
Locations (1):
- Ascension Genesys Hospital, Grand Blanc, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fong A, Serra AE, Caballero D, Garite TJ, Shrivastava VK. A randomized, double-blinded, controlled trial of the effects of fluid rate and/or presence of dextrose in intravenous fluids on the labor course of nulliparas. Am J Obstet Gynecol. 2017 Aug;217(2):208.e1-208.e7. doi: 10.1016/j.ajog.2017.03.010. Epub 2017 Mar 18. PMID 28322776
- [Background] Sharma C, Kalra J, Bagga R, Kumar P. A randomized controlled trial comparing parenteral normal saline with and without 5% dextrose on the course of labor in nulliparous women. Arch Gynecol Obstet. 2012 Dec;286(6):1425-30. doi: 10.1007/s00404-012-2485-1. Epub 2012 Aug 4. PMID 22865033
- [Background] ACOG Practice Bulletin No. 107: Induction of labor. Obstet Gynecol. 2009 Aug;114(2 Pt 1):386-397. doi: 10.1097/AOG.0b013e3181b48ef5. No abstract available. PMID 19623003
- [Background] Committee on Practice Bulletins-Obstetrics. Practice Bulletin No. 183: Postpartum Hemorrhage. Obstet Gynecol. 2017 Oct;130(4):e168-e186. doi: 10.1097/AOG.0000000000002351. PMID 28937571
- [Background] ACOG Committee Opinion No. 761: Cesarean Delivery on Maternal Request. Obstet Gynecol. 2019 Jan;133(1):e73-e77. doi: 10.1097/AOG.0000000000003006. PMID 30575678
- [Background] ACOG Committee Opinion No. 766: Approaches to Limit Intervention During Labor and Birth. Obstet Gynecol. 2019 Feb;133(2):e164-e173. doi: 10.1097/AOG.0000000000003074. PMID 30575638
- [Background] Philipson EH, Kalhan SC, Riha MM, Pimentel R. Effects of maternal glucose infusion on fetal acid-base status in human pregnancy. Am J Obstet Gynecol. 1987 Oct;157(4 Pt 1):866-73. doi: 10.1016/s0002-9378(87)80075-3. PMID 3314516
- [Background] Pare J, Pasquier JC, Lewin A, Fraser W, Bureau YA. Reduction of total labor length through the addition of parenteral dextrose solution in induction of labor in nulliparous: results of DEXTRONS prospective randomized controlled trial. Am J Obstet Gynecol. 2017 May;216(5):508.e1-508.e7. doi: 10.1016/j.ajog.2017.01.010. Epub 2017 Jan 30. PMID 28153654